CLINICAL TRIAL: NCT04186884
Title: Caregiver Burden, Quality of Life, and Symptom Distress at Different Palliative Cancer Care Settings
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2018-0819; NCI-2019-01197 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0819 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-03-28; First posted 2019-12-05 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Advanced Malignant Neoplasm; Locally Advanced Malignant Neoplasm; Metastatic Malignant Neoplasm; Recurrent Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaires): Patients and caregivers visiting SCC for a consult or admitted to PCU complete questionnaires over 35 minutes.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This trial studies caregiver burden, quality of life, and symptom distress of patients and their informal (unpaid) caregivers at different palliative care settings. Cancer caregiving may affect a caregiver's life physically, emotionally, socially, and financially. Studying caregiver burden may help investigators learn about caregivers' opinions on stress of caregiving, and about the factors related to caregiver burdens.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the severity of subjective stress burden (emotional impact) between caregivers of patients seen at the Supportive Care Center (SCC) and those seen at the Palliative Care Unit (PCU) as measured by the Montgomery - Borgatta Caregiver Burden Scale.

SECONDARY OBJECTIVES:

I. To compare objective burden (impact on tangible aspects of life) between caregivers of patients seen at SCC and the PCU.

II. To compare subjective demand burden (impact on the patient-caregiver relationship) between caregivers of patients seen at the SCC and the PCU.

III. To compare caregiver quality of life (measured by the Short-form 36) and symptom distress (measured by the caregiver ESAS [Edmonton Symptom Assessment System]) between caregivers of patients seen at the SCC and the PCU.

IV. To examine if there is a correlation between caregiver burden (Montgomery-Borgatta scale), quality of life (Short-form 36 scale) and symptom distress (ESAS caregiver scale).

V. To determine which caregiver and/or patients' factors are associated with caregiver burden, quality of life, and symptom distress.

OUTLINE:

Patients and caregivers visiting SCC for a consult or admitted to PCU complete questionnaires over 35 minutes.

ELIGIBILITY:
Inclusion Criteria

1. ( SCC Patient) Patients visiting the SCC for a first consultation.
2. (SCC Patient) Patients who can identify a primary informal caregiver.
3. (SCC Patient) Diagnosis of advanced cancer defined as locally advanced, recurrent, or metastatic.
4. (SCC Patient) Be able to read and speak English.
5. (SCC Patient) 18 years of age or older.
6. (Caregiver of SCC Patient) Be identified or self-identified as a primary informal caregiver of the patient. The caregiver could be present or verbally agree to participate.
7. (Caregiver of SCC Patient) Be able to read and speak English.
8. (Caregiver of SCC Patient) 18 years of age or older.
9. (Caregiver of SCC Patient) Caregivers who are not able to complete the assessment on the day of patients' first consultation must be willing to engage in a telephone assessment with research staff +/- 3 days after.
10. (PCU Patient) Patients who have been admitted to the PCU at MD Anderson Cancer Center.
11. (PCU Patient) Patients should have a primary informal caregiver during their PCU stay.
12. (PCU Patient) Diagnosis of advanced cancer defined as locally advanced, recurrent, or metastatic.
13. (PCU Patient) Be able to read and speak English.
14. (PCU Patient) 18 years of age or older.
15. (Caregiver of PCU Patient) Be identified by the patient or self-identified as the primary informal caregiver of the patient. The caregiver should be present with the patient during PCU stay.
16. (Caregiver of PCU Patient) Be able to read and speak English.
17. (Caregiver of PCU Patient) 18 years of age or older.

Exclusion Criteria

1. (SCC Patient) Refusal to participate in this study. This study requires both patient and caregiver enrollment.
2. (SCC Patient) Patients with only paid caregivers.
3. (SCC Patient) Patients with cognitive impairment as identified by research staff, treating physician or nurse.
4. (Caregiver of SCC Patient) Refusal to participate in this study. This study requires both patient and caregiver enrollment.
5. (Caregiver of SCC Patient) Patients with no caregivers or patients with only paid caregivers.
6. (PCU Patient) Refusal to participate in this study. This study requires both patient and caregiver enrollment.
7. (PCU Patient) Patients with no caregivers or patients with only paid caregivers.
8. (PCU Patient) Patients with cognitive impairment as identified by research staff, treating physician or nurse.
9. (Caregiver of PCU Patient) Refusal to participate in this study. This study requires both patient and caregiver enrollment.
10. (Caregiver of PCU Patient) Patients with no caregivers or patients with only paid caregivers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients visiting the SCC for a first consultation or patients admitted to the PCU at MD Anderson Cancer Center and primary informal caregiver of patient
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Severity of subjective stress burden (emotional impact) in caregivers of patients seen at the Supportive Care Center (SCC) and at the Palliative Care Unit (PCU) | Day 1, day of enrollment
  Measured by the Montgomery-Borgatta Caregiver Burden Scale. (4-item sub-scale questionnaire to measure the degree caregivers perceive their tasks and evaluates emotional effects of caregiving has a (Cronbach Alpha ranging from 0.68 to 0.82.)

SECONDARY OUTCOMES:
Objective burden (impact on tangible aspects of life Questionnaire | Day 1, day of enrollment
  Measured by Montgomery-Borgatta Caregiver Burden Scale using the 6-item objective burden sub-scale questionnaire. The sub-scale measure objective effects of caregiving in the caregivers life (i.e.:amount of time for personal privacy, recreational activities, time available to work, etc.) has a. Cronbach Alpha ranging from 0.87 to 0.90
Subjective demand burden (impact on the patient-caregiver relationship) of caregivers | Day 1, day of enrollment
  Measured by Montgomery-Borgatta Caregiver Burden Scale using the 4-item subjective demand burden sub-scale questionnaire. (ranges from 0.81 to 0.88)
Caregiver quality of life and symptoms of distress | Day 1, day of enrollment
  Will compare caregiver quality of life (measured by the Short-form 36) and caregiver symptom distress (measured by the caregiver Edmonton Symptom Assessment System [ESAS]) between caregivers of patients seen at the SCC and the PCU between caregivers of patients seen at the SCC and the PCU.(Cronbach Alpha ranges from 0.70 to 0.94)
Caregiver symptom distress | Day 1, day of enrollment
  Will examine the correlation between caregiver burden (Montgomery-Borgatta scale), quality of life (Short-form 36 scale) and symptom distress (ESAS caregiver scale). Explore if caregivers with higher burden will also have worse quality of life and higher symptom distress
Factors that are associated with caregiver burden, quality of life, and symptom distress Questionnaires | Day 1, day of enrollment
  Explore the effect of patients'caregivers' demographics, comorbidities (Charlson Comorbidity Index), duration of care since diagnosis, strength of religious faith and engagement (Santa Clara Strength of Religious Faith Questionnaire), trust in medical profession (Trust in the Medical Profession Questionnaire with caregiver burden, quality of life, patients' demographics and/or symptom distress, clinical characteristics (comorbidities, performance status, symptom distress scores, delirium severity prognosis) on each of caregivers' burden, quality of life, and symptom distress. Responses are summed and scores range from 5-25, with higher scores indicating higher trust

CONTACTS AND LOCATIONS:
Overall Officials: Kimberson C Tanco, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org